CLINICAL TRIAL: NCT00511147
Title: A Multi-center, Prospective, Open-label, Clinical Trial to Assess the Safety and the Efficacy of a New Intravenous Immune Globulin (IGIV3I Grifols 10%) in Patients With Idiopathic (Immune) Thrombocytopenic Purpura
Brief Title: IGIV Study for Chronic ITP Patients Ages 3-70
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grifols Biologicals, LLC (Industry)
Collaborators: Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IG0601
Record Dates: First submitted 2007-08-01; First posted 2007-08-03 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-05

CONDITIONS: Idiopathic Thrombocytopenic Purpura
Keywords: IVIG; ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IGIV3I Grifols 10% (All Subjects) (Experimental): All subjects with Chronic ITP
  Interventions: Biological: IGIV3I Grifols 10%

INTERVENTIONS:
Biological: IGIV3I Grifols 10% — IGIV3I Grifols 10% 1 g/kg/day given on two consecutive days, Day 1 and Day 2, for a total dose of 2 g/kg over two days.
  Other Names: Intravenous immunoglobulin

SUMMARY:
Idiopathic (immune) thrombocytopenic purpura (ITP) is an autoimmune disorder characterized by platelet destruction and thrombocytopenia (peripheral blood platelet count < 150 x 10^9/L). IVIG therapy is useful in patients in whom the platelet count has to be raised either due to bleeding signs, or where bleeding is predicted (e.g., surgery or parturition). The primary goal of treatment is to maintain the platelet count at a hemostatic level. This study will test the safety and efficacy of IGIV3I Grifols 10% in the treatment of patients with chronic ITP.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of chronic ITP
* Platelet count ≤ 20 x 10^9/L
* When administered corticosteroids at any time within 3 weeks before screening visit, the subject must have completed at least 3 weeks (21 days) of therapy at a stable and constant dose and schedule prior to screening visit
* When administered azathioprine (immunosuppressant) at any time within 3 months before screening visit, the subject must have received a stable dose and schedule for at least 3 months prior to screening visit
* When administered vinca alkaloids (eg., vincristine) at any time within 2 weeks before screening visit, the subject must have received a stable dose and schedule for at least 2 weeks prior to screening visit
* When administered attenuated androgens (eg, danazol) at any time within 8 weeks before screening visit, the subject must have received a stable dose and schedule for at least 8 weeks prior to screening visit.
* Females of childbearing potential must test negative for pregnancy

Key Exclusion Criteria:

* History or clinical evidence of medical conditions (other than ITP) felt to be the underlying cause of the thrombocytopenia
* Diagnosis of secondary immune thrombocytopenia
* History of severe (eg, anaphylactic) reactions to blood or any blood- derived product
* History of intolerance to any component of the IP, such as sorbitol
* Suffering serious and/or life-threatening hemorrhage/bleeding defined as:
* Any intracranial or central nervous system bleeding
* Any hemorrhagic event in which the subject is at risk of death at the time of the event
* Females who are pregnant or nursing an infant child
* Known to have immunoglobulin A (IgA) deficiency
* Known to abuse alcohol, opiates, psychotropic agents or other chemicals or drugs, or has done so within 12 months of the screening visit
* Documented diagnosis of thrombotic complications to polyclonal IVIG therapy in the past
* Unstable or uncontrolled disease, or condition, related to, or impacting, cardiac function: unstable angina, congestive heart failure, uncontrolled arterial hypertension
* Is anemic (hemoglobin < 9 g/dL)
* Renal impairment (ie, serum creatinine > 1.5 x upper limit of normal [ULN])
* Aspartate aminotransferase or alanine aminotransferase levels > 2.5 x ULN
* Known to have a positive test for either HCV or HIV (HIV 1/2)
* Splenectomy within the prior 8 weeks to the screening visit
* currently receiving any treatment for ITP except corticosteroids, azathioprine, vinca alkaloids or danazol
* Received an immune serum globulin (ISG) product within the prior 3 weeks (21 days) to the screening visit
* Received any alkylating agent (eg, cyclophosphamide) within 5 weeks prior to the screening visit
* Received rituximab within the prior 3 months to the screening visit
* Was currently receiving, or received, any therapeutic drug or device that was not approved by a Regulatory Authority (US or Canadian) for any indication within the prior 12 weeks to the screening visit

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Khojasteh, MD, Principal Investigator — Capitol Comprehensive Cancer Care Clinic
Locations (45):
- United States (31):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Scottsdale Medical Specialists, Scottsdale, Arizona
  - Arizona Oncology Associates, Tucson, Arizona
  - Scripps Cancer Center, La Jolla, California
  - Kenmar Research Institute, LLC, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Cancer Center of Central Connecticut, Southington, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - VA Medical Center, Washington D.C., District of Columbia
  - Halifax Health Medical Center, Daytona Beach, Florida
  - Hematology Oncology Associates, Lake Worth, Florida
  - Lakeland Regional Cancer Center, Tampa, Florida
  - St. Joseph's Children's Hospital of Tampa, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Emory University School of Medicine Winship Cancer Center, Atlanta, Georgia
  - Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Children's Hospital, New Orleans, Louisiana
  - Kalamazoo Hematology & Oncology, Kalamazoo, Michigan
  - CTO Breslin Cancer Center/MSU/Great Lakes Cancer Institute, Lansing, Michigan
  - University of Mississippi, Jackson, Mississippi
  - Capital Comprehensive Cancer Care Clinic, Jefferson City, Missouri
  - UMDNJ-RWJ Medical School, New Brunswick, New Jersey
  - Mt. Sinai Medical Center, New York, New York
  - Children's Hospital, University of Oklahoma, Oklahoma City, Oklahoma
  - Western Pennsylvannia Hospital, Pittsburgh, Pennsylvania
  - Baptist Cancer Center, Beaumont, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Tyler Hematology Oncology PA, Tyler, Texas
  - MCV Hospital, Richmond, Virginia
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - St. Joseph's Healthcare, Hamilton, Ontario
- India (11):
  - Narayana Hrudayalaya Hospitals, Karnataka, Bangalore
  - Shalby Hospitals, Ahmedabad
  - St. John's Medical College Hospital, Bangalore
  - Artemis Health Institute, Haryāna
  - Netaji Subhash Chandra Bose Cancer Research Institute, Kolkata
  - Christian Medical College, Ludhiana
  - Kodlikeri Hospital, Maharashtra
  - Grant Medical Foundation, Ruby Hall Clinic, Pune
  - Sahyadri Specialty Hospital, Pune
  - Apple Hospital, Surat
  - Christian Medical College, Vellore
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico

REFERENCES:
- [Derived] Apte S, Navarro-Puerto J, Damodar S, Ramanan V, John J, Kato G, Ross C, Shah C, Torres M, Fu C', Rucker K, Pinciaro P, Barrera G, Aragones ME, Ayguasanosa J. Safety and efficacy of intravenous immunoglobulin (Flebogamma(R) 10% DIF) in patients with immune thrombocytopenic purpura. Immunotherapy. 2019 Feb;11(2):81-89. doi: 10.2217/imt-2018-0165. Epub 2018 Nov 30. PMID 30499734

RESULTS

PARTICIPANT FLOW:
Groups:
- IGIV3I Grifols 10% (All Subjects): Intravenous immunoglobulin
  IGIV3I Grifols 10%: IGIV3I Grifols 10% 1 g/kg/day given on two consecutive days, Day 1 and Day 2, for a total dose of 2 g/kg over two days.
Period: Overall Study
Arm/Group | IGIV3I Grifols 10% (All Subjects)
Started | 64
Completed | 57
Not Completed | 7
Not completed — Withdrawal by Subject | 1
Not completed — Disease progression | 5
Not completed — Required platelet transfusion | 1

BASELINE CHARACTERISTICS:
Arm/Group | IGIV3I Grifols 10% (All Subjects)
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (18.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 32
  Black/African American | 2
  Hispanic/Latino | 6
  White | 24

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Defined by the percentage of treated patients in whom platelet counts increase from ≤ 20 x 10^9/L to ≥ 50 x 10^9/L by Day 8 ± 1 [where the day of the first infusion is Day 1]
Time Frame: 8 days
Population: Modified ITT Population
Measure: Number; unit: percentage of responders
Arm/Group | IGIV3I Grifols 10% (All Subjects)
Number analyzed (Participants) | 64
percentage of responders | 81.3

2. Secondary Outcome: Time to Platelet Count Recovery
Description: Defined by the number of days elapsed from Day 1 (the day of the first infusion of the IP) to the day when the platelet count is first known to be ≥ 50 x 10^9/L at any moment during the clinical follow-up period ending on Day 30 ± 1
Time Frame: 30 days
Population: Number of participants analyzed is based on the number of responding patients (52/64 [81.3%]) in the Modified ITT Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IGIV3I Grifols 10% (All Subjects)
Number analyzed (Participants) | 52
days | 1.7 (0.85)

3. Secondary Outcome: Duration of Response
Description: Defined by the number of consecutive days for which the platelet count remains ≥ 50 x 10^9/L at any moment during the clinical follow-up period ending on Day 30 ± 1.
Time Frame: 30 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IGIV3I Grifols 10% (All Subjects)
Number analyzed (Participants) | 52
days | 10.8 (7.69)

4. Secondary Outcome: Regression of Hemorrhage/Bleedings
Description: Defined by the percentage of treated patients with hemorrhage/bleedings at Day 1 (i.e., the day of the first infusion, pre-infusion) who improve their diathesis during the clinical follow-up period ending on Day 15 ± 1.
Time Frame: 15 days
Population: Number of participants analyzed is based on the number of patients with hemorrhage/bleeding at Day 1 in the Modified ITT Population
Measure: Number; unit: percent of subjects with regression
Arm/Group | IGIV3I Grifols 10% (All Subjects)
Number analyzed (Participants) | 44
percent of subjects with regression | 90.9

ADVERSE EVENTS:
Time Frame: 30 days follow-up
Arm/Group | IGIV3I Grifols 10% (All Subjects)
All-Cause Mortality (participants affected / at risk) | 0/64
Serious Adverse Events (participants affected / at risk) | 4/64
Other Adverse Events (participants affected / at risk) | 59/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IGIV3I Grifols 10% (All Subjects) (N=64)
meningitis aseptic (Infections and infestations) | 1
soft tissue inflammation (General disorders) | 1
Headache (Nervous system disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IGIV3I Grifols 10% (All Subjects) (N=64)
Nausea (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 9
Chills (General disorders) | 12
Pyrexia (General disorders) | 13
Body temperature increased (Investigations) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 7
Dizziness (Nervous system disorders) | 5
Headache (Nervous system disorders) | 41
Hypertension (Vascular disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 4
Contusion (Injury, poisoning and procedural complications) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Petechiae (Skin and subcutaneous tissue disorders) | 4
Hypotension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the study, after providing sponsor 30 days' notice prior to submitting a manuscript or other materials related to the study to any outside party. At sponsor's request, site will remove any confidential information (other than study results), and site will upon sponsor's request delay publication or presentation for a period of up to 120 days to allow sponsor to protect its interests in any sponsor inventions